CLINICAL TRIAL: NCT03755310
Title: Proof of Concept Study: Treatment of Restless Legs Syndrome With the Hypocretin Antagonist Suvorexant
Brief Title: Treatment of Restless Legs Syndrome With the Hypocretin Antagonist Suvorexant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diego García-Borreguero, MD, PhD (Other)
Collaborators: Sleep Research Institute (Paseo de la Habana 151, Madrid 28036, SPAIN) (Unknown)
Responsible Party: Sponsor-Investigator, Diego García-Borreguero, MD, PhD, Sleep Research Institute, Universidad Autonoma de Madrid
Organization: Universidad Autonoma de Madrid (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IISP-57325
Record Dates: First submitted 2018-08-10; First posted 2018-11-27 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Experimental): 10mg tabs during the first week, 10-20 mg tabs on the second week.
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Equivalent dosage, route of administration and dose regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — First week: 10 mg tabs; Second week: 10-20 mg tabs
  Arms: Suvorexant
Drug: Placebo — Equivalent dosage, route of administration and dose regimen
  Arms: Placebo

SUMMARY:
Suvorexant improves sleep latency and wake after sleep onset in patients with primary insomnia, and is FDA approved for this condition.

However, no data exist on its effects in RLS, so far. The investigators consider that suvorexant might provide a stable therapeutic efficacy for the long treatment, avoiding the risk of augmentation of symptoms commonly seen under dopamine agonists.

DETAILED DESCRIPTION:
Restless legs syndrome/Willis-Ekbom disease (RLS/WED) is a common neurological disorder characterized by the presence of an urge to move the legs, usually accompanied by dysesthesias1. It is estimated that approx. 60-75% of the patients experience these symptoms just at bedtime and its main consequence is insomnia. RLS is not only a common differential diagnosis with Primary Insomnia, but independently of this it is also one of the most common sleep disorders. In Western countries the prevalence for the more severe forms is approximately 2-3% of the general adult population.

Over the last years, dopamine agonists (DAs) have been widely used for RLS/WED. However, there is growing concern about the long-term consequences of DAs, such as dopaminergic augmentation. This complication consists of an overall increase in symptom severity, with symptoms starting earlier in the afternoon and expanding to previously unaffected parts of the body. If not stopped, augmentation can develop into a serious complication, as it will eventually progress and can lead to discontinuation of treatment. Existing studies show that after a treatment period of approximately 10 years, which is the amount of time that has elapsed since the first DA agonists were approved, the prevalence of augmentation nears 50%. But since RLS is a chronic disease in many patients, it is likely that with longer treatment times the risk of augmentation will increase even further. In light of this, there is a clinical need for treatment alternatives to dopaminergic drugs. Furthermore, a recent consensus paper by three RLS expert organizations recommends treatment begin with drugs other than dopaminergic agonists.

The pathophysiology of RLS/WED is not yet clear, but a number of findings link it to iron metabolism and to a mild dopaminergic dysfunction. Furthermore, it is not even clear whether the dopaminergic dysfunction plays a causal role at all, a fact that adds additional concerns about the use of dopaminergics. Drugs with non-dopaminergic mechanisms of action that have shown therapeutic efficacy for RLS/WED are alpha-2 delta ligands (pregabalin, gabapentin), opiates, benzodiazepines or clonidine. The only common mechanism through which these different agents might improve RLS symptoms is probably reduction of arousal. In fact, RLS even when moderate profoundly disturbs sleep, reducing sleep times to 5-6 hours or less. Patients report some daytime problems with alertness and cognitive clarity, but despite this reduction in sleep times untreated patients do not describe such profound episodes of sleepiness that occur for normal subjects maintained on such restricted sleep schedules. There is apparently some alerting mechanism partially compensating for the sleep loss. Such-hyperarousal-resembles the one found in Primary Insomnia. Indeed, RLS patients treated with dopaminergics over long periods frequently exhibit poor sleep despite the improvement of sensory and motor symptoms.

Increased glutamatergic activity has been discussed as one of the potential mechanisms leading to increased arousal in RLS. However, it is possible that the hypocretin system may also play a role in causing RLS-related hyperarousal. Hypocretins are well known to play a key role in the central regulation of both motor control and arousal. Two main studies have examined hypocretin levels in RLS patients. A first small study found increased evening hypocretin-1 levels in previously untreated patients with early onset RLS when compared to controls, but not in those treated. However, Stiasny-Kolster et al. were not able to replicate this finding, although the difference between both studies could be related to the treatment status and to the use of different extraction methods of cerebrospinal fluid (CSF). No evidence exists so far in the literature regarding the effect of hypocretin antagonist drugs in the treatment of RLS-related sensory and motor symptoms. However, unpublished data have shown non-significant improvements of periodic limb movements (PLMs) during treatment with almorexant.

This study hypothesizes that treatment of RLS symptoms with the hypocretin antagonist suvorexant might lead to an improvement of sleep as well as to an improvement of both dysesthesias and motor symptoms (PLMs).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic RLS, according to diagnostic criteria established by the International RLS Study Group (Allen et al., 2003).
* A history (if currently controlled on medication) or the presence of RLS symptoms causing insomnia/ sleep disturbance on 3 or more days per week for at least 12 months.
* Both treatment-naïve and treated patients without a sufficient response will be included. In both of these groups, the IRLS score ≥20 at the screening assessment (for the latter group, measured under current treatment), with an absence of significant RLS symptoms before 9PM (measured by diary)
* Aged 18 - 80 years.
* PSG at baseline containing:

  * WASO≥ 60 minutes
  * PLMAI of ≥ 15
  * TST<6.6hours
* Women of childbearing potential must have a negative pregnancy test at screen and must agree not to become pregnant.
* Prior to any study-specific procedures, a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Any secondary forms of RLS.
* History or current diagnosis of other clinically relevant diseases that may confound assessments or RLS symptoms.
* Serum ferritin <18 mcg/ml
* If the patient is currently being treated with drugs likely to influence sleep architecture or motor manifestations during sleep (such as neuroleptics, L-dopa, dopamine agonists, hypnotics, sedatives, antidepressants, anxiolytics, anticonvulsants, psychostimulant medications, steroids, barbiturates and opiates), a wash-out period of at least > 5 half-lives will be undertaken.
* Employed in shift work (for example, employment hours disruptive to the normal circadian sleep-wake cycle such as nighttime or variable rotating shifts) or irregular sleep-wake schedules.
* Patients who require prescription medication for concurrent conditions which could interfere with efficacy assessments such as dopamine antagonists, serotonin reuptake inhibitors or antihistamines.
* Surgery within 180 days of baseline visit, which in the opinion of the investigator would negatively impact the patient's participation in the study.
* A significant medical or psychiatric disorder.
* Any other clinically significant condition or laboratory assay abnormality, which would interfere with the patient's ability to participate in the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory assay abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and would make the patient inappropriate for entry into this study.
* Pregnancy and breastfeeding.
* Any disorders for which suvorexant is contraindicated, such as: narcolepsy, COPD, sleep apnea, depression, suicidal thoughts, severe hepatic illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change (differences between visits 2 and 5) in Wake Time After Sleep Onset (WASO), as measured during polysomnography | 1 year

SECONDARY OUTCOMES:
Change (differences between visits 2 and 5) in International Restless Legs Scale (IRLS) | 1 year
  IRLS is the main scale for rating the severity of restless legs syndrome. Scoring criteria: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40)
Change (differences between visits 2 and 5) in Clinical Global Impressions (CGI) | 1 year
Change (differences between visits 2 and 5) in Total Sleep Time (TST) | 1 year
Change (differences between visits 2 and 5) in Periodic Leg Movement during Sleep-index (PLMS) | 1 year
Change (differences between visits 2 and 5) in Periodic Leg movement while awake-index (PLMW-index) | 1 year
Change (differences between visits 2 and 5) in Multiple Suggested Immobilization Test (mSIT). | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Institute; Paseo de la Habana 151, Madrid, Spain

REFERENCES:
- [Background] 1. Sleep Med 2014;15(8):860-73. 2. Sleep Med. 2013;14(7):675-84. 3. Sleep Med 2012;13:1280-5. 4. Sleep Med 2011;12:440-4. 5. Sleep Med 2015;16(10):1252-8. 6. Sleep Med. 2016;21:1-11. 7. Sleep Med Clin 2015;10:207-14, xi. 8. Sleep Med. 2009;10(1):134-8. 9. Neurology. 2013;80(22):2028-34 10. Neurosci Biobehav Rev. 2015;49:43-54. 11. Peptides. 2014;52:29-37. 12. Curr Biol. 2013;23(18):1719-25. 13. Curr Opin Neurobiol. 2013;23(5):752-9. 14. Neurosci Bull. 2013;29(3):355-65. 15. Neurology. 2002;59(4):639-